CLINICAL TRIAL: NCT06694129
Title: Real-world Observational Study of Targeted Therapy in Patients With Advanced ROS1-positive NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Puyuan Xing, Chief Physician, National Cancer Center, China
Other Study IDs: NCC4601
Record Dates: First submitted 2024-11-03; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer; ROS1 Gene Rearrangement; Resistance; Targeted Therapy
Keywords: Non-Small Cell Lung Cancer; ROS1 Gene Rearrangement; Targeted therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — entrectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Tissue specimens or blood after resistance to entrectinib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: For eligible patients with advanced ROS1-positive NSCLC who have not received TKI treatment, receive entrectinib therapy until disease progression or intolerance.
  Interventions: Drug: Entrectinib
- Cohort 2: For patients with NSCLC who have progressed after receiving first-generation ROS1 TKI crizotinib and meet the eligibility criteria, they can receive entrectinib treatment until disease progression or intolerance.
  Interventions: Drug: Entrectinib
- Cohort 3: For patients with ROS1-positive NSCLC who have failed multi-line therapy, receive entrectinib until disease progression or intolerance.
  Interventions: Drug: Entrectinib

INTERVENTIONS:
Drug: Entrectinib — Patients in each cohort were treated with Entrectinib.
  Other Names: Rozlytrek

SUMMARY:
The purpose of this project is to conduct an observational study on the efficacy and safety of entrectinib in real-world patients with ROS1-positive NSCLC who have received entrectinib treatment, while exploring the mechanism of entrectinib's brain protection and resistance mechanism. Because this study is a non-interventional study, it will not interfere with your usual treatment. However, your medical data will be analyzed, and the results will help improve future treatment options for ROS1 positive NSCLC patients and improve their quality of life.This study was divided into three cohorts. Cohort 1: For patients with advanced ROS1-positive NSCLC who met the inclusion criteria and had not received TKI treatment, they were treated with entrectinib until disease progression or intolerance (N=15); Cohort 2: For patients with advanced ROS1-positive NSCLC who met the inclusion criteria and had received first-generation ROS1 TKI treatment with disease progression on crizotinib, they were treated with entrectinib until disease progression or intolerance (N=15); Cohort 3: For patients with ROS1-positive NSCLC who had failed multiple lines of treatment, they were treated with entrectinib until disease progression or intolerance (N=10). Regular follow-up was conducted and relevant clinical data were recorded, followed by Cox regression analysis and survival analysis. The information that needs to be recorded includes baseline and treatment genetic testing, demographic information, anti-cancer history, and concomitant medication use, as well as the use of study drugs and adverse events during treatment visits, survival and subsequent drug use after discharge, and the follow-up frequency consistent with clinical practice. Subjects are eligible for a complimentary NGS test upon the development of entrectinib resistance.

DETAILED DESCRIPTION:
The purpose of this project is to conduct an observational study on the efficacy and safety of entrectinib in real-world patients with ROS1-positive NSCLC who have received entrectinib treatment, while exploring the mechanism of entrectinib's brain protection and resistance mechanism. Because this study is a non-interventional study, it will not interfere with your usual treatment. However, your medical data will be analyzed, and the results will help improve future treatment options for ROS1 positive NSCLC patients and improve their quality of life.This study was divided into three cohorts. Cohort 1: For patients with advanced ROS1-positive NSCLC who met the inclusion criteria and had not received TKI treatment, they were treated with entrectinib until disease progression or intolerance (N=15); Cohort 2: For patients with advanced ROS1-positive NSCLC who met the inclusion criteria and had received first-generation ROS1 TKI treatment with disease progression on crizotinib, they were treated with entrectinib until disease progression or intolerance (N=15); Cohort 3: For patients with ROS1-positive NSCLC who had failed multiple lines of treatment, they were treated with entrectinib until disease progression or intolerance (N=10). Regular follow-up was conducted and relevant clinical data were recorded, followed by Cox regression analysis and survival analysis. The information that needs to be recorded includes baseline and treatment genetic testing, demographic information, anti-cancer history, and concomitant medication use, as well as the use of study drugs and adverse events during treatment visits, survival and subsequent drug use after discharge, and the follow-up frequency consistent with clinical practice. Subjects are eligible for a complimentary NGS test upon the development of entrectinib resistance.

ELIGIBILITY:
Inclusion Criteria:

* 1) Histologically or cytologically confirmed non-small cell lung cancer;
* 2) TNM stage of the ninth edition is IIIB, IIIC, or IV;
* 3) ROS1 fusion positive confirmed by one of the following qualified results: next-generation sequencing technology, fluorescence in situ hybridization, reverse transcription polymerase chain reaction;
* 4) No prior systemic chemotherapy, radiation therapy, or surgery;
* 5) Aged 18 years or older;
* 6) ECOG PS score of 0-1.

Exclusion Criteria:

* 1) any prior history of NSCLC and/or any prior treatment for NSCLC;
* 2) prior systemic chemotherapy or radiation therapy or surgical treatment;
* 3) the presence of a second primary tumor;
* 4) hypersensitivity to ROS1-TKI or intolerance to it.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-small cell lung cancer exhibiting ROS1 rearrangement.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From enrollment to the end of treatment at 1 year.

SECONDARY OUTCOMES:
Objective remission rate | From enrollment to the end of treatment at 1 year.
Time to CNS progression | From enrollment to the end of treatment at 1 year.
Overall survival | From enrollment to the end of treatment at 1 year.

OTHER OUTCOMES:
Exploratory biomarker analysis | From enrollment to the end of treatment at 1 year.

IPD SHARING:
Plan to Share IPD: No
It involves patient privacy and cannot be disclosed at will.